CLINICAL TRIAL: NCT01065675
Title: Electronic Patient Triage Development and Implementation Involving Nurse (RN), Pharmacy Technician (CPhT), and Pharmacist (RPh) Obtained Medication Histories in the Emergency Department (ED)and Impact on Medication Reconciliation
Brief Title: Medication Histories Conducted by Nurses (RNs), Pharmacy Techs (CPhTs) & Pharmacists (RPhs)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Statistical analysis of 153 enrolled Phase 1 patients showed that specific patients could not be targeted for medication histories by discipline.
Sponsor: Wesley Medical Center (Other)
Collaborators: Cardinal Health (Industry)
Responsible Party: Principal Investigator, Joan Kramer, Clinical Research Pharmacist, Wesley Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: 09-068
Record Dates: First submitted 2010-02-03; First posted 2010-02-09 (Estimated); Last update posted 2012-12-28 (Estimated); Status verified 2012-12

CONDITIONS: Medication Reconciliation; Emergency Department
Keywords: Medication Reconciliation; Emergency Department; Nurse; Pharmacist; Certified Pharmacy Technician; Medication reconciliation: inpatients admitted from the ED
MeSH Terms: conditions — Emergencies | interventions — Medication Reconciliation; Pharmacists; Nurses; Emergency Service, Hospital

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Medication reconciliation completed by a RN, CPhT, or RPh — To determine which patients benefit the most from medication histories obtained by the RN, CPhT, or RPh. Patients will be admitted as inpatients through the ED with medication histories finalized electronically by the RN at the admitting unit.
  Other Names: Medication Reconciliation; Pharmacist; Nurse; Certified Pharmacy Technician; Emergency Department; ED

SUMMARY:
Up to 50% of medication errors and 20% of adverse drug reactions (ADRs) in the hospital setting are estimated to be related to communication issues regarding patient medications at various transition points of care from admission to discharge. The Joint Commission (TJC) requires accurate and complete medication reconciliation occur at each transition point throughout hospitalization. Evidence from NQF demonstrates pharmacists (RPh) are the most effective medication management team leaders in the implementation of medication management practices and design of medication error reduction strategies; medication reconciliation is one of the five safety objectives pharmacists are recommended to lead. In addition, the Massachusetts Coalition for the Prevention of Medical Errors states strong evidence supports the use of pharmacy technicians (CPhT) in conjunction with pharmacists in completing accurate medication histories.

WMC nurses (RN) currently are involved in the medication reconciliation process. In 2009, a Medication Use Evaluation (MUE) of Medication Reconciliation Accuracy found a 67% medication error rate on admission determined by comparing the nurse-obtained medication history to the pharmacist-obtained medication history. The number of home medications identified by the pharmacist compared to the nurse was 411 versus 312 (p<0.0001). The total percentage of medication errors prevented by the pharmacist was 66.2. Using the VA Healthcare Failure Mode Effects Analysis - HFMEA™ Hazard Scoring Matrix, 3 independent pharmacist reviewers found that 18% of patients interviewed had a score greater than 7, and 3 patients had a score of 12 (major/probable), if the discrepancies would not have been identified and corrected by the pharmacist conducting the admission medication reconciliation audit. The same patients' discharge medication reconciliation and discharge medication lists were retrospectively reviewed for the MUE, and the total percentage of patients with medication errors on discharge was 43%.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted as inpatients from the Emergency Department

Exclusion Criteria:

* Prisoners (because the IRB does not have a prisoner representative)
* Patients not admitted as inpatients through the Emergency Department
* Patients admitted more than once during the study period

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2010-02; Primary Completion 2010-04 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
To determine which patients benefit most from medication histories obtained by the RN, CPhT, or RPh based on accuracy (% complete disease states, allergy documentation and description, vaccination documentation, medication documentation) | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Joan S Kramer, PharmD, Principal Investigator — Wesley Medical Center
Locations (1):
- Wesley Medical Center, Wichita, Kansas, United States